CLINICAL TRIAL: NCT00811369
Title: A Phase II, Multi-Centre, Randomized, Double-blind Trial to Evaluate the Therapeutic Benefit of Fulvestrant in Combination With ZACTIMA or Fulvestrant Plus Placebo in Postmenopausal Women With Bone Only or Bone Predominant, Hormone Receptor Positive Metastatic Breast Cancer
Brief Title: Trial to Evaluate the Therapeutic Benefit of Fulvestrant in Combination With ZACTIMA in Postmenopausal Women With Bone Predominant, Hormone Receptor Positive Metastatic Breast Cancer
Acronym: ZAMBONEY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OCOG-2008-ZAMBONEY
Record Dates: First submitted 2008-12-15; First posted 2008-12-19 (Estimated); Last update posted 2013-11-18 (Estimated); Status verified 2013-11

CONDITIONS: Metastatic Breast Cancer
Keywords: Breast Cancer; Bone Metastases; Telopeptide; Zactima; Fulvestrant
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant; vandetanib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Fulvestrant + ZACTIMA Group
  Interventions: Drug: Fulvestrant + ZACTIMA
- 2 (Placebo Comparator): Fulvestrant + Placebo Group
  Interventions: Drug: Fulvestrant + Placebo

INTERVENTIONS:
Drug: Fulvestrant + ZACTIMA — ZACTIMA 100 mg tablets. Dose = 1 tablet daily until disease progression or intolerance
  Other Names: Vandetanib
  Arms: 1
Drug: Fulvestrant + Placebo — ZACTIMA Placebo 100 mg tablets. Dose = 1 tablet daily for duration of study.
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate whether the combination of fulvestrant and ZACTIMA, versus fulvestrant plus placebo, results in a significant decrease in the bone marker, urinary N-Telopeptide (NTx) in postmenopausal women with bone only, or bone predominant, hormone receptor-positive metastatic breast cancer. A significant decrease will be defined as a > 30% reduction in urinary NTx level from baseline.

DETAILED DESCRIPTION:
Tumor angiogenesis is associated with invasiveness and the metastatic potential of various cancers. Vascular endothelial growth factor (VEGF), the most potent and specific angiogenic factor, regulates normal and pathologic angiogenesis. The increased expression of VEGF has been correlated with metastases, recurrence and poor prognosis in many cancers. It has been shown the VEGF is involved in osteolysis in women with bone metastases. ZACTIMA is an agent which targets VEGF. ZACTIMA is a new agent with novel method of action - it is a VEGF inhibitor, epidermal growth factor (EGFR) inhibitor, tyrosine kinase inhibitor, as well as a potential RET kinase activity inhibitor.

In summary, women with bone only, or bone predominant, metastatic breast cancer is an ideal group to study anti-angiogenic therapies where angiogenesis could be a major factor in tumor progression and where anti-angiogenic treatment with agents like ZACTIMA could be more effective.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal woman, defined as a woman fulfilling any one of the following criteria:

   * Age greater than or equal to 60 years or
   * Age greater than or equal to 45 years with amenorrhea more than 12 months with an intact uterus or
   * Follicle-stimulating hormone (FSH) levels in postmenopausal range or
   * Having undergone a bilateral oophorectomy
2. Metastatic breast cancer with either radiologically confirmed bone only or predominant metastases to bone not considered amenable to curative treatment.
3. Evidence of hormone sensitivity either ER+ and/or PgR+, as per institutional standards, in the primary tumor.
4. Patients must fulfill one of the following RECIST criteria:

   * Bone lesions, which are lytic, sclerotic or mixed (lytic + sclerotic), in the absence of measurable disease as defined by RECIST criteria or
   * Bone lesions, which are lytic, sclerotic or mixed (lytic + sclerotic), in the presence of measurable disease as defined by RECIST criteria.
5. Patients must fulfill one of the following resistances to endocrine therapy criteria:

   * Disease progression on tamoxifen or on an aromatase inhibitor as first or second line therapy for metastatic disease or
   * Development of metastatic disease while on treatment with tamoxifen or an aromatase inhibitor in the adjuvant setting or
   * Disease progression after discontinuation of prior adjuvant endocrine therapy.

Exclusion Criteria:

1. Previous treatment with fulvestrant or ZACTIMA.
2. History of hypersensitivity to active or inactive excipients of fulvestrant and/or ZACTIMA.
3. Has received greater than one line of systemic chemotherapy for metastatic breast cancer.
4. Has received chemotherapy within the past 14 days (+ 2 days).
5. Has received radiation therapy within the past 14 days (+ 2 days).
6. Has undergone major surgery within the past 21 days or has had major surgery performed > 21 days prior to screening and the wound remains unhealed.
7. Has received LH-RH agonist within the past 4 months.
8. Prior treatment with VEGF inhibitors (prior use of AVASTIN permitted).
9. Current or previously active systemic malignancy within 3 years prior to randomization (other than breast cancer, or adequately treated in-situ carcinoma of the cervix, uteri, or basal or squamous cell carcinoma of the skin).
10. Presence of life-threatening metastatic visceral disease, defined as extensive hepatic involvement, or any degree of brain or leptomeningeal involvement (past or present), or symptomatic pulmonary lymphangetic spread. Patients with discrete pulmonary parenchymal metastases are eligible, provided their respiratory function is not compromised as a result of disease.
11. ECOG performance status of > 2.
12. Currently receiving (and are unwilling to discontinue) hormone replacement therapy.
13. Laboratory results sustained at:

    * Platelets < 100 x 109 /L
    * International normalized ratio (INR) > 1.6
    * Total bilirubin > 1.5 times normal
    * ALT or AST > 2.5 times normal range if no demonstrable liver metastases or > 5 times normal range in the presence of liver metastases. No more than three retests within screening period are allowable.
14. Potassium level outside of normal range, despite supplementation; serum calcium (or ionized or adjusted for albumin), or magnesium below the lower limit of the normal range despite supplementation or creatinine clearance < 30mL/min.
15. History of:

    * Bleeding diathesis (i.e. disseminated intravascular coagulation [DIC], clotting factor deficiency) or
    * Long-term anticoagulant therapy (other than anti-platelet therapy).
16. Any severe concomitant condition which makes it undesirable for the patient to participate in the study or which would jeopardize compliance with the protocol, e.g. severe renal or hepatic impairment or currently unstable or uncompensated respiratory or cardiac conditions, ongoing or active infection, untreated primary hyperparathyroidism, or psychiatric illness that would limit compliance with study requirements.
17. Anticipated life expectancy less than six months.
18. Non-approved/experimental drug treatment within previous 4 weeks before randomization.
19. Significant cardiovascular event (e.g., myocardial infarction, superior vena cava syndrome), New York Heart Association (NYHA) classification of heart disease (Appendix II) > Class II within 3 months before study entry, or presence of cardiac disease that in the opinion of the investigator increases the risk of ventricular arrhythmia.
20. History of arrhythmia (multifocal premature ventricular contractions (PVCs), bigeminy, trigeminy, ventricular tachycardia, or uncontrolled atrial fibrillation) which is symptomatic or requires treatment (NCI CTCAE Grade 3 or 4) or asymptomatic sustained ventricular tachycardia. Atrial fibrillation, controlled on medication, is not excluded.
21. Congenital long QT syndrome or 1st degree relative with unexplained sudden death under 40 years of age.
22. QT prolongation with other medications that required discontinuation of that medication.
23. Presence of left bundle branch block (LBBB).
24. QTc with Bazett's correction measurable at > 480msec on screening ECG. (Note: If a patient has QTc > 480msec on screening ECG, the screen ECG may be repeated twice (at least 24 hours apart). The average QTc from the three screening ECGs must be < 480msec in order for the patient to be eligible for the study). Patients who are receiving a drug that has a risk of QTc prolongation (see Appendix III, Table 2) are excluded if QTc is > 460msec.
25. Hypertension not controlled by medical therapy (systolic blood pressure > 160 millimeter of mercury (mmHg) or diastolic blood pressure > 100mmHg).
26. Concomitant medications that are potent inducers (rifampicin, rifabutin, phenytoin, carbamazepine, phenobarbital and St. John's Wort) of CYP3A4 function.
27. Not accessible for treatment and follow up.
28. Failure to provide informed consent.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2009-08; Primary Completion 2012-10 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Significant change in NTx level defined as a ≥ 30% reduction in urinary NTx level from baseline. | Week # 1-4, 12, and every 12 weeks until disease progression/recurrence

SECONDARY OUTCOMES:
Progression free survival (PFS) | Every 12 weeks until disease progression/recurrence
Response to therapy | Every 12 weeks until disease progression/recurrence
Improvement in pain | Week # 1-4, 12, and every 12 weeks until disease progression/recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Mark Clemons, MD, Principal Investigator — The Ottawa Hospital Regional Cancer Centre; Rebecca Dent, MD, Principal Investigator — Odette Cancer Centre - Sunnybrook Health Sciences Centre
Locations (13):
- Canada (13):
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency - Vancouver Centre, Vancouver, British Columbia
  - QE II Health Sciences Centre, Halifax, Nova Scotia
  - Regional Cancer Program of the Hôpital régional de Sudbury Regional Hospital, Greater Sudbury, Ontario
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Grand River Regional Cancer Centre, Kitchener, Ontario
  - RSM Durham Regional Cancer Centre, Oshawa, Ontario
  - Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Odette Cancer Centre - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Centre Hospitalier De L'Universite De Montreal - Hotel Dieu, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan